CLINICAL TRIAL: NCT06508931
Title: A Single-arm, Multi-center, Open-label Phase II Study to Determine the Safety and Efficacy of MB-CART2019.1 in Pediatric Subjects With Relapsed/Refractory Mature B-cell Neoplasms Who Have Relapsed After One or More Prior Therapies, Including Subjects With Primary Refractory Disease
Brief Title: Safety and Efficacy Study of Zamtocabtagene Autoleucel (MB-CART2019.1) in Pediatric Patients With R/R B-Cell Neoplasms
Acronym: DALY PED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Collaborators: PPD, Part of Thermo Fisher Scientific (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2021-389; 2023-506348-17-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-02; First posted 2024-07-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: B-Cell Neoplasm
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: A multi-center, international, open-label study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- zamtocabtagene autoleucel (MB-CART2019.1) (Experimental)
  Interventions: Drug: zamtocabtagene autoleucel (MB-CART2019.1)

INTERVENTIONS:
Drug: zamtocabtagene autoleucel (MB-CART2019.1) — Tandem CD20-CD19-directed non-cryopreserved CAR-T cell therapy.

SUMMARY:
This is a single-arm, multi-center, open-label Phase II study to determine the safety and efficacy of MB-CART2019.1 in pediatric and adolescent subjects (aged between 6 months and <18 years, ≥6 kg body weight [BW]) with mature B-cell neoplasms and aggressive lymphomas that relapsed after or are refractory to one or more prior therapies, including subjects with primary refractory disease.

DETAILED DESCRIPTION:
This is a single-arm, multi-center, open-label Phase II study designed to evaluate the efficacy of zamtocabtagene autoleucel (MB-CART2019.1) therapy infusion in pediatric subjects with relapsed/refractory (r/r) mature B-cell neoplasms. The primary study endpoint will be best overall response (BORR). Furthermore, the safety and toxicity of the study product will be assessed based on type, frequency, and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESI).

MB-CART2019.1 is designed to effectively target malignant B cells in patients suffering from haematological B-cell malignancies. Zamtocabtagene autoleucel (MB-CART2019.1) is a tandem CD20-CD19-directed non-cryopreserved CAR-T cell therapy. Pediatric patients who are suitable for this study will be treated with MB-CART2019.1.

Zamtocabtagene autoleucel (MB-CART2019.1) administration consists of a single infusion with fresh formulation of 2.5 × 10^6 CAR-transduced autologous T cells/kg bodyweight. IMP is only to be administered after a lymphodepleting chemotherapy with fludarabine and cyclophosphamide. For MB-CART2019.1 production, pediatric patients will undergo a leukapheresis. The enrollment period will last approximately 36 months and the duration of the study for each subject will be 85 weeks (including screening period and a 78 weeks safety follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Is able to provide age-appropriate assent/consent (as applicable, according to local legislation) and/or have a guardian able to provide consent signed and dated by the parent(s) or by subject's legal guardian before conduct of any study-specific procedures.
2. Has histologically confirmed mature CD19+ and/or CD20+ B-cell neoplasm such as:

   * Burkitt lymphoma/Burkitt leukemia
   * Diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS)
   * Primary mediastinal (thymic) large B-cell lymphoma
   * Burkitt-like lymphoma with 11q aberration
   * Aggressive mature B-cell lymphoma
   * Other rare aggressive B-cell non-Hodgkin lymphoma (NHL) after sponsor approval.
3. Has r/r B-cell neoplasms after one or more prior therapies or primary refractory to first-line therapy.
4. Is a pediatric/adolescent (aged between 6 months and <18 years).
5. Has a BW of ≥ 6 kg.
6. Measurable disease based on the International Pediatric NHL Response Criteria (which refers to the Lugano criteria for definitions of measurability and selecting index lesions), as identified by local radiological assessment for lymphomas. Previously irradiated lesions cannot be considered measurable unless the lesion has proven radiological evidence for progression after the radiation.
7. Tissue samples archival or fresh (preferred) from recent relapse or initial diagnosis (in case of primary refractory disease) must be made available for the central pathology review to confirm diagnosis (≤2 years, preferably not older than 2 months since collection).
8. Has Karnofsky (aged ≥16 years) or Lansky (aged <16 years) performance status ≥60.
9. Has adequate bone marrow function as defined by the following laboratory values (as assessed by local laboratory for eligibility):

   * Absolute neutrophil count (ANC) >1000/μL.
   * Platelets ≥50000/μL.
   * Hemoglobin ≥8.0 g/dL.
   * Absolute lymphocyte count ≥100/μL.
10. Has adequate organ function as follows:

    * Renal function: estimated glomerular filtration rate (eGFR) >29 mL/min by Schwartz formula (Schwartz et al 1976).
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 × upper limit of normal (ULN) for age.
    * Bilirubin <1.5 x ULN (for Gilbert's Syndrome, subject's total bilirubin <4 mg/dL).
    * Adequate pulmonary function as follows:

      * Resting oxygen saturation of ≥91% on room air.
      * No or mild dyspnea (Grade ≤1).
11. Female subjects of childbearing potential must be willing to undergo pregnancy tests before MB-CART2019.1 infusion.
12. If subjects are sexually active, they must be willing to use highly effective methods of contraception.

    * Female subjects must agree to use two methods of contraception;

      * one of the following methods (Pearl index <1%): Hormonal contraceptives associated with inhibition of ovulation (oral, intravaginal, injected, implanted, transdermal), intrauterine devices (IUDs) or systems (e.g., hormonal and non-hormonal IUD), or vasectomized sexual partner AND one barrier method.
      * Highly effective methods of contraception must be followed from inclusion until 12 months after MB-CART2019.1 infusion.
    * Male subjects must agree to use a condom during intercourse from inclusion through at least 12 months after MB-CART2019.1 infusion to prevent them from fathering a child AND to prevent delivery of MB-CART2019.1 via seminal fluid to their partner. Do not use a female condom when using a male condom, since tearing can occur. In addition, male subjects must not donate sperm for the time period specified above.
    * Females must agree not to breast feed or donate eggs/ova during the study and until at least 12 months after MB-CART2019.1 infusion.
13. Is willing to undergo collection of non-mobilized leukapheresis.
14. In the opinion of the investigator, the subject must be able to comply with all study-related procedures, medication use, and assessments.

Exclusion Criteria:

1. Is receiving active treatment for malignant disease (including participation in any additional parallel investigational drug or device studies), except for pre-enrollment therapy, including radiotherapy. Lesions that are irradiated during pre-enrollment therapy may not be considered measurable lesions. For subjects with lymphoma to be eligible, there must be at least one measurable lesion after pre-enrollment therapy.
2. Had allogeneic HSCT.
3. Had autologous HSCT <120 days prior to written informed consent.
4. Had major surgery within 2 weeks before leukapheresis, or has not fully recovered from an earlier surgery, or has major surgery planned during the time the subject is expected to participate in the study.
5. Subjects with B-cell neoplasms in the context of post-transplant lymphoproliferative disorders-associated lymphomas.
6. Has known hypersensitivity to the excipients of the MB-CART2019.1 or to any other drug product as advised for administration in the study protocol (e.g., lymphodepleting agents).
7. Has active central nervous system (CNS) involvement at the time point of eligibility confirmation, as measured by the presence of lymphoma cells in cerebral spinal fluid (CSF) on cytospin preparation.
8. Has history or presence of autoimmune CNS disease, such as multiple sclerosis, optic neuritis, or other immunologic or inflammatory diseases.
9. Infection with human immunodeficiency virus (HIV).
10. Presence of active or prior hepatitis B or C as indicated by serology. Treated infection with hepatitis B or C virus unless confirmed to be polymerase chain reaction (PCR) negative.
11. Has infection with Treponema pallidum.
12. Has active infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
13. Has infection with human T-lymphotropic virus 1/2 (HTLV 1/2).
14. Has active severe systemic fungal, viral, or bacterial infection, requiring systemic antiviral, antifungal, or antimicrobial therapy.
15. Has clinically significant seizures according to the opinion of by the investigator.
16. Has history of cerebral vascular accident within 12 months prior to leukapheresis.
17. Has impaired cardiac function: Fractional shortening <28% or left ventricular ejection fraction <50% by echocardiography or multigated acquisition, if allowed as per local law.
18. Has concomitant genetic syndromes associated with bone marrow (BM) failure status, such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known BM failure syndrome.
19. Is a pregnant or breast-feeding female.
20. Is sexually active and not willing to use highly effective methods of contraception as described in the inclusion criteria.
21. Has history of another malignancy within the prior 3 years that required systemic therapy.
22. Has other medical, psychological, or social condition that, in the opinion of the investigator, would impact subject safety or confound the study results.
23. Has received vaccination with live virus within 6 weeks prior to informed consent.
24. Has been previously treated with approved anti-CD19 or anti-CD20 CART cell therapies <100 days prior to informed consent/assent.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
BORR, Best Overall Response Rate | From infusion until week 78
  The primary efficacy outcome of this study is BORR, defined as the proportion of subjects with at least one partial response (PR) or complete response (CR) from MB-CART2019.1 infusion until progressive disease (PD), start of new anti-lymphoma therapy, lost to follow-up or death, whichever occurs first.
Type, frequency, and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESI) [Safety and toxicity of the study product] | From infusion until week 78
  The primary safety outcome of this study is to evaluate the incidence, type, frequency, and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESI) associated with the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Burkhardt, Prof. Dr., Principal Investigator — Uniklinik Münster, Klinik für Kinder- und Jugendmedizin Pädiatrische Hämatologie/Onkologie
Locations (1):
- Institut Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No